CLINICAL TRIAL: NCT03272217
Title: A Phase II Trial of Atezolizumab and Bevacizumab in Cisplatin-ineligible Patients With Advanced/Unresectable Urothelial Cancer
Brief Title: Atezolizumab With Bevacizumab in Previously Untreated Metastatic/Unresectable Urothelial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funder decision
Sponsor: Arjun Balar, MD (Other)
Collaborators: Roche-Genentech (Industry); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Arjun Balar, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU15-215; NCT03133390 (obsolete NCT alias)
Record Dates: First submitted 2017-09-01; First posted 2017-09-05 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Urothelial Carcinoma
Keywords: Atezolizumab; MPDL3280A; Bevacizumab; Avastin; Cisplatin-Ineligible; Anti-PD-L1 Antibodies
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm A - Atezolizumab + Bevacizumab (Experimental): Patients will receive atezolizumab 1200 mg (flat dose) IV plus bevacizumab 15 mg/kg IV every 21 days
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg (flat dose) IV every 21 days
  Other Names: MPDL3280A
Drug: Bevacizumab — Bevacizumab 15 mg/kg IV every 21 days
  Other Names: Avastin

SUMMARY:
This is a phase II study assessing the activity of bevacizumab combined with atezolizumab in metastatic urothelial carcinoma patients who are ineligible for cisplatin-based therapy.

DETAILED DESCRIPTION:
This is a multi-center trial.

INVESTIGATIONAL TREATMENT:

Eligible patients will be receive atezolizumab 1200 mg IV flat dose plus bevacizumab 15 mg/kg IV every 21 days

21 days equals 1 cycle of therapy and patients will be eligible to continue treatment until progressive disease by RECIST v1.1 or unacceptable toxicity for up to 24 months.

To demonstrate adequate organ function, all screening labs must be obtained within 14 days prior to Cycle 1 Day 1 (C1D1) of treatment:

Hematological:

* Absolute Neutrophil Count (ANC): ≥ 1,000 K/mm^3
* Hemoglobin (Hgb): ≥ 9.0 g/dL
* Absolute Lymphocyte Count: ≥ 500/uL
* Platelet Count: ≥ 100,000/uL

Renal:

* Calculated Creatinine Clearance: serum creatinine < 2.5 or ≥ 25 cc/min using a direct method or the Cockcroft-Gault formula
* Urinary Protein Excretion: < 1.0 g/24 hours (as estimated by urine protein-creatinine ratio)

Hepatic:

* Bilirubin: ≤ 1.5 × upper limit of normal (ULN) (patients with known Gilbert's Disease who have serum bilirubin ≤ 3.0 x ULN may be enrolled)
* Aspartate aminotransferase (AST): ≤ 2.5 × ULN (5.0 x ULN if liver involvement)
* Alanine aminotransferase (ALT): ≤ 2.5 × ULN (5.0 x ULN if liver involvement)
* Serum Albumin: ≥ 2.5 g/dL

Coagulation:

* International Normalized Ratio (INR) or Prothrombin Time (PT); Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 × ULN (NOTE: This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose)

ELIGIBILITY:
INCLUSION CRITERIA

Patient must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization for release of personal health information.
* As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with study procedures for the entire length of the study
* Age ≥ 18 years at the time of consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2 within 28 days prior to registration
* Histological or cytological evidence urothelial (transitional cell) carcinoma of the renal pelvis, ureter, bladder or urethra
* Locally advanced/unresectable disease as determined by site attending urologic oncologist or metastatic disease
* Evaluable untreated tumor tissue for biomarker analysis. Untreated tumor tissue is defined as no intervening intravesical or systemic therapy since acquisition. Patients without tissue available must be willing and safe to undergo biopsy repeat biopsy (core needle or excisional) prior to enrollment. Subjects with < 25 slides may be enrolled after discussion with the sponsor-investigator or co-investigator.
* Willing to undergo a core needle or excisional biopsy on-treatment. Patients will be assessed at the time of biopsy for safety of undergoing the procedure
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 within 28 days prior to registration
* No prior chemotherapy for locally advanced or metastatic urothelial cancer

  * Perioperative chemotherapy previously administered in the neoadjuvant and/or adjuvant setting is permitted
  * Prior chemotherapy administered in the context of chemoradiation as definitive treatment for bladder preservation is also permitted, provided that disease progression outside the prior radiotherapy field is demonstrated histologically or cytologically
* Ineligible for cisplatin as defined by presence of one or more of the following:

  * (Impaired renal function [≤ 60 cc/min]. Glomerular filtration rate (GFR) should be assessed by direct measurement [i.e., creatinine clearance or ethylenediaminetetra-acetate] or, if not available, by calculation from serum/plasma creatinine by Cockroft-Gault equation)
  * Grade ≥ 2 hearing Loss (measured by loss of >25 dB at two contiguous frequencies in at least one ear for patients undergoing serial audiometry testing)
  * Grade ≥ 2 peripheral neuropathy
  * ECOG Performance Status of 2
  * Solitary Kidney
  * Refusing Cisplatin-based chemotherapy
* If palliative radiotherapy administered, completion of palliative radiation therapy ≥ 2 weeks prior to Cycle 1 Day 1 of protocol therapy
* Females of childbearing potential must have a negative serum pregnancy test within 28 days prior to registration.
* Females of childbearing potential and males must be willing to abstain from heterosexual intercourse or to use 2 forms of effective methods of contraception from the time of informed consent until 150 days (5 months) after discontinuation of atezolizumab or 180 days (6 months) after discontinuation of bevacizumab. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method

EXCLUSION CRITERIA

Patients meeting any of the criteria below may not participate in the study:

* Any approved anti-cancer therapy, including chemotherapy, or hormonal therapy within 3 weeks prior to initiation of study treatment; the following exceptions are allowed:

  * Palliative radiotherapy for bone metastases or soft tissue lesions should be completed > 7 days prior to baseline imaging
  * Hormone-replacement therapy or oral contraceptives
* Treatment with any other investigational agent or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment
* Active or untreated central nervous system (CNS) metastases or leptomeningeal disease as determined by computed tomography (CT) scan or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments.
* Patients with treated asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

  * Evaluable or measurable disease outside the CNS
  * No metastases to midbrain, pons, medulla, cerebellum, or within 10 mm of the optic apparatus (optic nerves and chiasm)
  * No history of intracranial or spinal cord hemorrhage
  * No evidence of significant vasogenic edema
  * No ongoing requirement for dexamethasone as therapy for CNS disease; anticonvulsants at a stable dose allowed
  * No stereotactic radiation, whole-brain radiation within 4 weeks prior to Cycle 1 Day 1
  * Patients with central nervous system (CNS) metastases treated by neurosurgical resection or brain biopsy within 3 months prior to Cycle 1 Day 1 will be excluded
  * Radiographic demonstration of interim stability (i.e., no progression) between the completion of CNS-directed therapy and the screening radiographic study
  * Screening CNS radiographic study ≥ 4 weeks since completion of radiotherapy or surgical resection and ≥ 2 weeks since discontinuation of corticosteroids
* Leptomeningeal disease
* Uncontrolled tumor-related pain

  * Patients requiring pain medication must be on a stable regimen at study entry
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

  * Patients with indwelling drainage catheters are allowed.
* Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or Ca > 12 mg/dL or corrected serum calcium > ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab. NOTE: Patients with asymptomatic hypercalcemia controlled with medical therapy are eligible.

  * Patients who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.
  * Patients who are receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate instead while in the study.
* Malignancies other than urothelial cancer within 5 years prior to Cycle 1 Day 1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, or ductal carcinoma in situ treated surgically with curative intent) or localized prostate cancer treated with curative intent and absence of prostate-specific antigen (PSA) relapse or incidental prostate cancer (T1/T2a, Gleason score ≤ 3 + 4, and PSA ≤ 0.5 ng/mL undergoing active surveillance and treatment naive)
* Pregnant or breastfeeding
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab or bevacizumab formulation
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, granulomatosis with polyangiitis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis

  * Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
  * Subjects with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
  * Subjects with a history of celiac disease may be eligible if controlled with diet.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* History of confirmed positive test for human immunodeficiency virus (HIV)
* Patients with active hepatitis B virus (HBV) (chronic or acute, defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C virus (HCV)

  * Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* Active tuberculosis
* Severe infections within 4 weeks prior to Cycle 1 Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of active infection within 2 weeks prior to C1D1
* Received therapeutic oral or IV antibiotics within 1 week prior to C1D1

  * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible
* New York Heart Association Congestive Heart Failure Class II or greater
* Myocardial infarction, unstable angina or unstable arrhythmias within 3 months of enrollment.
* History of stroke or TIA within 3 months of enrollment
* Other clinically significant arterial vascular disease within 6 months of enrollment (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis). Prior history of adequately treated venous thromboembolism > 7 days prior to C1D1 on stable dose of therapeutic anticoagulation is permitted
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Major surgical procedure other than for diagnosis within 28 days prior to C1D1 or anticipation of need for a major surgical procedure during the course of the study
* Prior allogeneic stem cell or solid organ transplant
* Administration of a live, attenuated vaccine within 4 weeks before C1D1 or anticipation that such a live attenuated vaccine will be required during the study
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications

ATEZOLIZUMAB-SPECIFIC EXCLUSION CRITERIA:

* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies

  * Prior cancer vaccines and cellular immunotherapy are permitted.
* Treatment with systemic immunostimulatory agents (including but not limited to IFNs, interleukin [IL]-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to C1D1
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to C1D1, or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids, physiologic replacement doses of glucocorticoids (i.e., for adrenal insufficiency), and mineralocorticoids (e.g., fludrocortisone for adrenal insufficiency) is allowed

BEVACIZUMAB-SPECIFIC EXCLUSION CRITERIA:

* Inadequately controlled hypertension (defined as persistent systolic blood pressure (SBP) > 150 and/or diastolic blood pressure (DBP) > 100 mmHg)
* Prior history of hypertensive crisis or hypertensive encephalopathy
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study enrollment) use of aspirin (> 325 mg/day), clopidogrel (> 75 mg/day), or current or recent (within 10 days prior to first dose of bevacizumab) use of therapeutic oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes
* History of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment
* Minor surgical procedure within 7 calendar days prior to C1D1
* History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to enrollment
* Clinical signs or symptoms of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious non-healing or dehiscing wound, active ulcer, or untreated or non-healing bone fracture
* On-going gross hematuria associated with clots

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-13 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2022-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Balar, M.D., Study Chair — Hoosier Cancer Research Network
Locations (8):
- United States (8):
  - University of Arizona at Dignity Health St. Joseph, Phoenix, Arizona
  - Rush University Medical Center, Chicago, Illinois
  - HealthPartners Institute, Minneapolis, Minnesota
  - New York University Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - West Cancer Center University of Tennessee, Memphis, Tennessee
  - Froedtert & The Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 77 [54 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate at 1 Year
Description: Determine the percentage of overall survival at 1 years from the initiation of treatment. Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: 1 years
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 16
Percentage of participants | 67

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter(LD) of target lesions; Progressive Disease (PD): >= 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
  Overall Response (OR) = CR + PR.
Time Frame: Up to a maximum of 14 months
Population: Out of 16 subjects, one had no response. Therefore 15 subjects were evaluable for ORR.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 15
Percentage of participants | 6.67

3. Secondary Outcome: Duration of Response (DOR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  DOR is defined as time from measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented by RECIST v1.1.
Time Frame: Up to a maximum of 14 months
Population: Only one subject achieve complete or partial response by RECIST v1.1.
Measure: Number; unit: Months
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 1
Months | 6.54

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time from the date of treatment start until the criteria for disease progression is met as defined by RECIST 1.1 or death occurs
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 36 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 16
Months | 3.25 [2.07 to NA] — Upper limit was not reached due to an insufficient number of participants with events.

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events were recorded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.
Time Frame: Adverse events were recorded from time of registration until 30 days after discontinuation of study drug(s), up to maximum of 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Atezolizumab + Bevacizumab
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 36 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 12 months.
Arm/Group | Arm A - Atezolizumab + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 6/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Atezolizumab + Bevacizumab (N=16)
ANEMIA (Blood and lymphatic system disorders) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
FEVER (General disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PAIN (General disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 2 (2)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (3)
WOUND INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Atezolizumab + Bevacizumab (N=16)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 (5)
AGITATION (Psychiatric disorders) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (5)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ANEMIA (Blood and lymphatic system disorders) | 9 (19)
ANOREXIA (Metabolism and nutrition disorders) | 4 (8)
ASCITES (Gastrointestinal disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
AUTOIMMUNE DISORDER (Immune system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
BLADDER SPASM (Renal and urinary disorders) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (2)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CHEST PAIN - CARDIAC (Cardiac disorders) | 1 (1)
CHILLS (General disorders) | 5 (7)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 (1)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 3 (4)
CONSTIPATION (Gastrointestinal disorders) | 4 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE INCREASED (Investigations) | 7 (10)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 2 (3)
DIZZINESS (Nervous system disorders) | 2 (4)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DUODENAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 3 (3)
EDEMA LIMBS (General disorders) | 3 (6)
EYE DISORDERS - OTHER, SPECIFY (Eye disorders) | 1 (1)
FACIAL PAIN (General disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 9 (9)
FEVER (General disorders) | 5 (15)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 (5)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
FLU LIKE SYMPTOMS (General disorders) | 1 (2)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 (8)
HEADACHE (Nervous system disorders) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 2 (4)
HEMOGLOBINURIA (Renal and urinary disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 6 (12)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPONATREMIA (Metabolism and nutrition disorders) | 4 (12)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 3 (4)
HYPOTHYROIDISM (Endocrine disorders) | 2 (2)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
IMMUNE SYSTEM DISORDERS - OTHER, SPECIFY (Immune system disorders) | 1 (1)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (3)
INSOMNIA (Psychiatric disorders) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (1)
LYMPHEDEMA (Vascular disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (1)
MUCOSAL INFECTION (Infections and infestations) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 3 (3)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 2 (4)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 4 (7)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 2 (3)
PROTEINURIA (Renal and urinary disorders) | 5 (11)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (6)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (2)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 2 (4)
RENAL COLIC (Renal and urinary disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 3 (3)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 2 (4)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (3)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY FREQUENCY (Renal and urinary disorders) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 4 (6)
URINARY TRACT OBSTRUCTION (Renal and urinary disorders) | 1 (3)
URINARY TRACT PAIN (Renal and urinary disorders) | 2 (2)
VASCULAR DISORDERS - OTHER, SPECIFY (Vascular disorders) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 4 (6)
WEIGHT LOSS (Investigations) | 3 (4)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03272217/Prot_SAP_000.pdf